CLINICAL TRIAL: NCT01686022
Title: The Study of Allergens From Grass and Weed Which Are Causes of Allergic Rhinitis in Thai Patients
Brief Title: Grass Sensitisation and Allergic Rhinitis in Thai Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Punchama Pacharn, Principal investigator, Mahidol University
Other Study IDs: NRCT_G04
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Allergy to Grass Pollen; Allergic Rhinitis Due to Weed Pollens
Keywords: Grass; Major allergen; cross-reactivity
MeSH Terms: interventions — Immunoblotting

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pollen Allergy: Pollen allergy and control will have the same intervention, ie. Skin prick test and collect serum samples.Then measure the specificIgE, immunoblot, and ELISA inhibition
  Interventions: Other: Immunoblot

INTERVENTIONS:
Other: Immunoblot — serum specific IgE binds to grass extract by immunoblot

SUMMARY:
Allergic rhinitis patients are the patients who have nasal symptoms when triggered by indoor or outdoor allergens. Outdoor allergen can be divided into grass, tree, or weed. The type of grass or weed are different in various part of the world. The allergens from grass and weed has never been studied in Thailand. This study will find the major allergen from Bermuda grass, Johnson grass, Para grass, sedge, and ragweed, which are very common in Thailand. In addition, the investigators will study about the cross-reactivity among these group of allergen.

DETAILED DESCRIPTION:
To find the major allergen of grass and weed, the serum of patients will be used to bind with the allergen extract by immunoblot study.

The ELISA-inhibition will be used to study about cross-reactivity among various kinds of grass and weed.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis patients age 10-50 years old
* Control: healthy volunteer age 18-50 years old

Exclusion Criteria:

* Chronic illness such as cardiovascular diseases, liver diseases
* History of anaphylaxis
* Pregnancy

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Allergy Clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided